CLINICAL TRIAL: NCT00935506
Title: Evaluation of an Experimental EX Vivo Thrombosis Chamber Model in Healthy Male Subjects
Brief Title: Ex Vivo Human Thrombosis Chamber Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CV197-004
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2010-04

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clopidogrel + Aspirin (Experimental)
  Interventions: Drug: Clopidogrel; Drug: Aspirin

INTERVENTIONS:
Drug: Clopidogrel — Tablets, Oral, 75 mg, Once daily, 8 days
  Other Names: Plavix
Drug: Aspirin — Tablets, Oral, 325 mg, Once daily, 8 days

SUMMARY:
Purpose of study is to evaluate a thrombosis chamber model

ELIGIBILITY:
Inclusion Criteria:

* Healthy Subjects
* BMI 18-30 kg/m²
* Male ages 18-45

Exclusion Criteria:

* Significant acute or chronic illness
* History of abnormal bleeding or coagulation disorder, intracranial hemorrhage, or a family history of abnormal bleeding or coagulation disorder in a first degree relative under 50 years of age
* Easy bruising
* Smoking within 3 months prior to Day 1

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2009-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Evaluate ex vivo thrombosis chamber model by assessing the effect of anti-platelet agents on thrombus formation | Period 2, Day 8

SECONDARY OUTCOMES:
Assess variability of thrombosis chamber measurements | Period 1 and Period 2
Assess relationship between platelet aggregation and thrombus formation | Period 1 and Period 2
Safety and tolerability of multiple doses clopidogrel and aspirin | From Day 1 through Study Discharge

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Mds Pharma Services, Neptune City, New Jersey, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx